CLINICAL TRIAL: NCT04884113
Title: PowerSpiral Enteroscopy: Multicenter Prospective Study on Performance and Safety Including Patients With Altered Gastrointestinal Anatomy
Brief Title: PowerSpiral Enteroscopy Performance and Safety
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Abdulbaqi Al-Toma, Principal investigator, St. Antonius Hospital
Other Study IDs: W20.204
Record Dates: First submitted 2021-05-03; First posted 2021-05-12 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Small Bowel Disease
Keywords: Motorized Spiral enteroscopy; Device-assisted enteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Motorized Spiral Enteroscopy: Procedure: Motorized Spiral Enteroscopy:
  PowerSpiral enteroscope will be inserted and advanced with the assistance of motorized spiral rotation, After reaching the point of maximum insertion, cecum or if no further advancement of the enteroscope can be achieved, the enteroscope will be withdrawn using motorized counter-clockwise spiral rotation. When no total enteroscopy is reached, submucosal ink dye injection is performed as an endoscopically visible marker of the maximum insertion depth. A retrograde enteroscopy is then performed in the same session or at second session
  Interventions: Device: Motorized Spiral enteroscopy

INTERVENTIONS:
Device: Motorized Spiral enteroscopy — Small-bowel enteroscopy for diagnosis and intervention

SUMMARY:
Multicenter study to evaluate the efficacy of the motorized spiral enteroscope in the management of small bowel diseases.

DETAILED DESCRIPTION:
Background and Aims:

Motorized Spiral enteroscopy is a recent advancement in enteroscopy. Data are scarce on the utility and safety of the motorized spiral enteroscopy. No data is available on the utility of this technique in patients with altered gastrointestinal (GI) anatomy.

This study aimed to evaluate the efficacy of motorized spiral enteroscopy including rate of total enteroscopy (TER) in patients undergoing enteroscopy for suspected small bowel disease including those with altered GI anatomy.

Methods: A multicenter prospective study evaluated consecutive patients with symptomatic small bowel disease who underwent enteroscopy over a 12-month period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Patients with suspected small bowel pathology indicated for diagnostic and/or therapeutic enteroscopy based on clinical presentation, small bowel imaging, or video capsule enteroscopy
3. Written informed consent

Exclusion Criteria:

1. Contraindications for endoscopy because of comorbidities
2. Unable to provide written informed consent
3. Patients with known severe gastrointestinal tract inflammation, intestinal obstruction, gastroesophageal varices or eosinophilic esophagitis that preclude a safe enteroscopy procedure
4. Coagulopathy or thrombocytopenia that could not be corrected by blood product transfusion
5. Pregnant patients
6. Health status: American Society of Anesthesiologists (ASA) class >3
7. Inability to tolerate Propofol sedation or general anesthesia for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected small bowel pathology indicated for diagnostic and/or therapeutic enteroscopy based on clinical presentation, small bowel imaging, or video capsule enteroscopy
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
The diagnostic yield of motorized spiral enteroscopy | 2 days
  Diagnostic yield achieved by antegrade and/or retrograde enteroscopy using motorized spiral enteroscopy
The therapeutic yield of motorized spiral enteroscopy | 2 days
  Total number of therapeutic interventions performed during antegrade and/or retrograde enteroscopy using the motorized spiral enteroscopy

SECONDARY OUTCOMES:
Total enteroscopy rate | 2 days
  Estimate the number of total enteroscopy procedures achieved by either antegrade only or antegrade and retrograde motorized spiral enteroscopy
Technical success | 2 days
  Estimate the rate of technically successful enteroscopy procedures both antegrade and retrograde motorized spiral enteroscopy
Total procedural time | 2 days
  The total time needed to complete the whole procedure of enteroscopy antegrade and/or retrograde motorized spiral enteroscopy
Depth of maximum insertion into the small bowel | 2 days
  Estimation of the maximum depth of insertion (in centimeters) both antegrade and/or retrograde motorized spiral enteroscopy
Adverse events | 7 days
  Total minor and also serious adverse events during and after antegrade and/or retrograde motorized spiral enteroscopy

CONTACTS AND LOCATIONS:
Overall Officials: A Al-Toma, Ph.D., Principal Investigator — St. Antonius Hospital
Locations (5):
- Netherlands (5):
  - VU University Medical Center, Amsterdam
  - University Medical Centre Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - Maastricht UMC+, Maastricht
  - St Antonius hospital, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Toma A, Beaumont H, Koornstra JJ, van Boeckel P, Hergelink DO, van der Kraan J, Inderson A, de Ridder R, Jacobs M. The performance and safety of motorized spiral enteroscopy, including in patients with surgically altered gastrointestinal anatomy: a multicenter prospective study. Endoscopy. 2022 Nov;54(11):1034-1042. doi: 10.1055/a-1783-4802. Epub 2022 Feb 28. PMID 35226945